CLINICAL TRIAL: NCT01758822
Title: Role of Endotracheal Suction on the Occurrence of Meconium Aspiration Syndrome in Non-vigorous Meconium Stained Neonates- A Randomized Controlled Trial
Brief Title: Role of Endotracheal Suction on the Occurrence of Meconium Aspiration Syndrome in Non-vigorous Meconium Stained Babies
Acronym: ETMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Professor of Pediatrics, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHMC/2011/PED/019
Record Dates: First submitted 2012-12-20; First posted 2013-01-01 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Meconium Aspiration Syndrome
Keywords: meconium stained amniotic fluid; endotracheal suction; non vigorous neonates
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Endotracheal suction (Experimental): In the experimental group, endotracheal suction will not be performed during the initial steps of resuscitation of non-vigorous meconium stained neonate
  Interventions: Other: No endotracheal suction
- Endotracheal suction (No Intervention): In the No intervention group endotracheal suction will be performed during the initial steps of resuscitation of non - vigorous meconium stained neonate

INTERVENTIONS:
Other: No endotracheal suction — Neonates in this group will be resuscitated without endotracheal suction in the initial steps of resuscitation.
  Arms: No Endotracheal suction

SUMMARY:
The purpose of this study is to evaluate the role of endotracheal suction on the occurrence of meconium aspiration syndrome in depressed meconium stained babies. Meconium aspiration syndrome (MAS) is believed to result from aspiration of meconium and consequent chemical pneumonitis. Meconium can be aspirated into the lungs in the womb as well. Meconium in the distal airways is not accessible to endotracheal (ET) suction which clears only the windpipe. Furthermore there is growing evidence in support of asphyxia-hypoxia-acidosis in the causation of lung disease. Moreover, in the absence of a clear role of ET suction in depressed meconium stained newborns, critical time could be lost in assessment, intubation and ET suction (range: 30 seconds to 1 min) which might delay the definitive step of ventilation for resuscitation of such babies that can potentially affect the outcome adversely.The utility or futility of endotracheal suction in preventing MAS in depressed meconium stained neonates has not been systematically studied and there is inadequate information in literature in favor or against this practice.Thus this study is an attempt to evaluate the effect of endotracheal suction on the occurrence of MAS in depressed full term neonates born through meconium stained amniotic fluid (MSAF).

DETAILED DESCRIPTION:
Approximately 10-15% of deliveries are complicated by the passage of meconium around the time of delivery.An adverse intrauterine environment with resultant fetal asphyxia is proposed as the most common explanation for in-utero passage of meconium.

Aspiration of meconium into the tracheo-bronchial tree with the onset of respiration results in meconium aspiration syndrome (MAS). MAS is defined as respiratory distress in an infant born through MSAF with compatible chest x-ray findings whose symptoms cannot be otherwise explained.

Despite current interventions such as intubation and tracheal suction, it is estimated that 5-20 % of infants born through MSAF develop MAS. It represents a leading cause of perinatal morbidity. Approximately 50% of the infants with MAS require mechanical ventilation; 15%-30% develop pulmonary air leaks and 5%-12% die.

There are various proposed mechanisms by which meconium causes lung injury, some of the important ones being

* Mechanical obstruction of airways
* Chemical pneumonitis
* Vasoconstriction of pulmonary vessels
* Inactivation of surfactant
* Activation of compliment

Finding of meconium below cords or in the trachea has been shown to be associated with development of MAS. This resulted in use of endotracheal suction along with oro-nasopharyngeal suctioning in all infants born to mothers with MSAF prior to the year 2000.

Although, a number of studies performed did not show reduction in incidence of MAS and/or mortality even after performing oro-nasopharyngeal and endotracheal suction, the practice was continued due to lack of robust evidence.

Subsequently, as a result of well performed randomized controlled trials and systematic review showing no effect of oro-nasopharyngeal suctioning on occurrence of MAS, this practice has been abandoned since the year 2005.

ET suction is currently performed in depressed meconium stained neonates with the idea of removing meconium from the upper airways to relieve mechanical obstruction and to prevent subsequent development of chemical pneumonitis.

Since meconium aspiration can occur in-utero as well and with time the aspirated meconium migrates peripherally, the effectiveness of ET suction post-delivery in clearing the airway is not clear. Furthermore, accumulating evidence points to potential role of hypoxia-asphyxia-acidosis with concomitant presence of meconium in the pathogenesis of lung disease.

Current practice of Endotracheal suctioning in non-vigorous babies has not been systematically evaluated, till date. No studies have compared the incidence, severity and outcomes of MAS in 'suctioned versus non-suctioned' non vigorous meconium stained neonates. In addition, the procedure needs expertise to be completed in the stipulated time and has potential for complications like vocal cord injury, laryngeal edema, bleeding from upper airway secondary to trauma during the procedure and persistent hoarseness of voice even at six months of age. The rate of complications is more when performed by people with lesser expertise as this is a difficult skill to learn and master.

In view of the foregoing the contribution of endotracheal suction in preventing MAS and its effect on severity of lung disease is not clear. Thus this study is an attempt to evaluate the role of endotracheal suction in non-vigorous meconium stained neonates.

ELIGIBILITY:
Inclusion Criteria:

* Gestation age > 37 weeks
* Cephalic Presentation
* Singleton pregnancy
* Presence of meconium stained amniotic fluid
* Nonvigorous at birth

Exclusion Criteria:

* Major congenital malformations
* Refusal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of MAS and death due to all cause | till discharge or death up to 6 weeks of life
  MAS is defined as meconium staining of liquor or staining of nails or umbilical cord or skin along with presence of any one of the following:
  * Respiratory distress within one hour of birth OR
  * Radiological evidence of aspiration pneumonitis (atelectasis and/or hyperinflation)

SECONDARY OUTCOMES:
Duration of oxygen therapy | till discharge or death up to 6 weeks of life
  duration of oxygen therapy in hours
Duration and severity of respiratory distress by Downe's scoring | till discharge or death up to 6 weeks of life
  Severity of respiratory distress is assessed using Downe's score, the parameters are documented hourly within first twelve hours and then every two hourly till persistence of respiratory distress for first seventy hours( whichever is shorter) and on four hourly basis after seventy hours in the presence of respiratory distress.
Need for and duration of Mechanical ventilation in hours | Till discharge or death up to 6 weeks of life
  Total duration of mechanical ventilation, mode and ventilator parameters noted till the baby is on ventilator
HIE(hypoxic ischemic encephalopathy) staging | During the first two weeks of life
  by Sarnat and Sarnat classification system
Incidence of complications | till death or discharge up to 6 weeks of life
  incidence of PPHN, pneumothorax suspected on clinical basis and confirmed by echocardiography and chest radiography respectively and incidence of sepsis
Duration of hospital stay | till death or discharge up to 6 weeks of life
  duration of hospital stay in completed days

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MBBS, MD, DM, Principal Investigator — Lady Hardinge Medical College New Delhi, India
Locations (1):
- Kalawati Saran children's Hospital, Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Nangia S, Sunder S, Biswas R, Saili A. Endotracheal suction in term non vigorous meconium stained neonates-A pilot study. Resuscitation. 2016 Aug;105:79-84. doi: 10.1016/j.resuscitation.2016.05.015. Epub 2016 May 30. PMID 27255954